CLINICAL TRIAL: NCT00592930
Title: Pilot Study of the Efficacy of Olanzapine in the Treatment of Anorexias Nervosa
Brief Title: Olanzapine in the Treatment of Anorexia Nervosa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Vivian Kafantaris, M. D., North Shore- Long Island Jewish Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 99-04-072; Lilly F1D-US-X166
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2008-01-14 (Estimated); Status verified 2008-01

CONDITIONS: Anorexia Nervosa
Keywords: anorexia nervosa, treatment, adolescents, olanzapine
MeSH Terms: conditions — Anorexia Nervosa | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): olanzapine
  Interventions: Drug: olanzapine
- 2 (Placebo Comparator): matching placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: olanzapine — flexibly dosed oral olanzapine 2.5 to 15 mg/day
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
This study compared 10 weeks of treatment with olanzapine versus placebo in adolescent females with anorexia nervosa-restricting type who were undergoing acute treatment on an inpatient unit or a day hospital program that specializes in the treatment of eating disorders.

ELIGIBILITY:
Inclusion Criteria:

* Females, ages 12-23

Exclusion Criteria:

* Binge-purge type

Ages: 12 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20
Dates: Start 2000-06; Primary Completion 2004-12 (Actual); Study Completion 2004-12

PRIMARY OUTCOMES:
weight gain | 10 weeks

SECONDARY OUTCOMES:
measures of psychiatric symptoms | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Kafantaris, M.D., Principal Investigator — Schneider Children's Hospital
Locations (1):
- Schneider Children's Hospital, New Hyde Park, New York, United States

REFERENCES:
- [Derived] Kafantaris V, Leigh E, Hertz S, Berest A, Schebendach J, Sterling WM, Saito E, Sunday S, Higdon C, Golden NH, Malhotra AK. A placebo-controlled pilot study of adjunctive olanzapine for adolescents with anorexia nervosa. J Child Adolesc Psychopharmacol. 2011 Jun;21(3):207-12. doi: 10.1089/cap.2010.0139. PMID 21663423